CLINICAL TRIAL: NCT05093062
Title: Efficacy Observation on Tian Jiu Therapy for Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: HHSRF 12133081
Record Dates: First submitted 2019-02-27; First posted 2021-10-26 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tian Jiu Therapy (Other)
  Interventions: Other: Tian Jiu Therapy

INTERVENTIONS:
Other: Tian Jiu Therapy

SUMMARY:
Objectives:

To further evaluate the immediate, long-term and cumulative effects of Tian Jiu Therapy on asthma.

Hypothesis to be tested:

The efficacy of Tian Jiu Therapy on asthma is also long-term and will be accumulated.

Design and Subjects:

Recruiting 167 asthma participants who received Tian Jiu Therapy under the primary study of HKCTR-1128. All subjects should be above age 13 and receive the same Tian Jiu Therapy, 3 times per year from 2013 to 2015. A one-year follow-up after the last Tian Jiu treatment will be conducted.

Study instruments:

Modern USB PC-based Spirometer and Fingertip Pulse Oximeter.

Interventions:

Plastering some stimulating Chinese herbal cubes on certain acupoints in the three hottest days of each year, for three consecutive years.

Main outcome measures:

Pulmonary Function Test, Blood Oxygen Test, Quality of Life and Standardized Questionnaire on asthma attack and symptoms will be administered before treatment, after treatment of each year and one-year follow-up after the last treatment.

Data analysis:

All the parameters will be analyzed, the physical improvement (Cured, Remarkably effective, Effective and Ineffective) will be recorded, and the differences in different treatment courses will be investigated and compared with previous data obtained in the primary study of HKCTR-1128 by using standard statistical analysis.

Expected results:

The effect of Tian Jiu Therapy on Asthma is not only immediate but also long-term and will be gradually accumulated.

The Tian Jiu Therapy will acquire better efficacy on asthma if this treatment was conducted more years continuously.

ELIGIBILITY:
Inclusion Criteria:

- History of Asthma

Diagnostic Criteria of Asthma according to U.S.DHHS(2007):

1. Episodic symptoms of airflow obstruction
2. Difficulty breathing
3. Chest tightness
4. Cough (worse at night)
5. Symptoms occurring or worsening at night, awakening the patient
6. Symptoms occurring or worsening with exercise, viral infections, changes in weather, strong emotions, or mens; or in the presence of animals, dust mites, mold, smoke, pollen, or chemicals
7. Wheezing
8. Airflow obstruction at least partially reversible Medically stable and acute medical care does not require. E.g. intensive monitoring, invasive ventilation, haemoid-dialysis, cardiac support.

Exclusion Criteria:

1. Patients currently experiencing Acute asthma attack
2. Infants and child under thirteen years old 3.Pregnant women

4. Patients with

1. Fever and pharyngitis
2. Tuberculosis
3. Severe cardiac and pulmonary diseases
4. Diabetes Mellitus
5. Hypersensitive skin condition
6. Allergy to topical medication
7. Keloid
8. Bleeding disorders
9. Severe heart diseases and with pacemaker.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
The change in Quality of life | baseline, change from baseline at 1-2th week; change from baseline at 12 months after treatment
  The change in Quality of life (SF-36 score)
The change in the frequency of asthma attack | baseline, change from baseline at 1-2th week; change from baseline at 12 months after treatment
  The change in the frequency of asthma attack
The change in admission to hospital | baseline, change from baseline at 1-2th week; change from baseline at 12 months after treatment
  The change in admission to hospital
The change in AE visit | baseline, change from baseline at 1-2th week; change from baseline at 12 months after treatment
  The change in AE visit
The change in clinic visit | baseline, change from baseline at 1-2th week; change from baseline at 12 months after treatment
  The change in clinic visit

SECONDARY OUTCOMES:
The change of Pulmonary Function (FEV1) | baseline, change from baseline at 1-2th week; change from baseline at 12 months after treatment
  The change of Pulmonary Function (FEV1)
The change of Pulmonary Function (FEV1/FEC) | baseline, change from baseline at 1-2th week; change from baseline at 12 months after treatment
  The change of Pulmonary Function (FEV1/FEC)